CLINICAL TRIAL: NCT03221816
Title: Effect of Polyvitaminics (Pyridoxine Hydrochloride, Folic Acid and Cyanocobalamin) in the Concentration of Homocysteine and Lipid Profile in Postmenopausal Women: a Randomized Controlled, Double-blind Clinical Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Casa de Saúde santa Marcelina (Other)
Responsible Party: Principal Investigator, Carolina Vicente Banzoli, Principal Investigator, Casa de Saúde santa Marcelina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: U1111-1176-6998
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Menopause; Dyslipidemias; Homocystinaemia
Keywords: Menopause; homocysteine; lipid profile
MeSH Terms: conditions — Dyslipidemias | interventions — Pyridoxine; Folic Acid; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Oral Tablet (Placebo Comparator): Sixty women were postmenopausal selected from the outpatient Gynecology Hospital Santa Marcelina that passed by routine consultations and fulfilling the inclusion criteria were invited to the study.
  The women were randomly allocated to control or experimental group (30 in each group) in a double-blind controlled clinical trial.
  The control group received the same tablet with the organoleptic characteristics of Tenavit® for a period of 4 months.
  Interventions: Drug: Placebo Oral Tablet
- Experimental group (Tenavit®) (Experimental): Sixty women were postmenopausal selected from the outpatient Gynecology Hospital Santa Marcelina that passed by routine consultations and fulfilling the inclusion criteria were invited to the study.
  The experimental group received one tablet of Tenavit® (pyridoxine hydrochloride 4.00mg + folic acid 0.80mg + cyanocobalamin 0.40 mg) daily and the placebo group received the same tablet with the organoleptic characteristics of Tenavit® for a period of 4 months.
  Interventions: Drug: Tenavit®

INTERVENTIONS:
Drug: Tenavit® — The experimental group received one tablet of Tenavit® daily for a period of 4 months.
  Other Names: pyridoxine, folic acid, cyanocobalamin
  Arms: Experimental group (Tenavit®)
Drug: Placebo Oral Tablet — Placebo group received the same tablet with the organoleptic characteristics of Tenavit® for a period of 4 months.
  Other Names: Placebo
  Arms: Placebo Oral Tablet

SUMMARY:
Introduction: Cardiovascular diseases (CVD) are the main cause of death in Western countries. High levels of homocysteine (He) has been considered an important risk factor for coronary artery disease. Objective: To evaluate the effects of the drug Tenavit® (pyridoxine hydrochloride 4.00mg + folic acid 0.80mg + cyanocobalamin 0.40 mg) on plasma homocysteine concentrations and lipid profile in postmenopausal women. Methods: Sixty women were postmenopausal selected from the outpatient Gynecology Hospital Santa Marcelina that passed by routine consultations and fulfilling the inclusion criteria were invited to the study. The women were randomly allocated to control or experimental group (30 in each group) in a do uble-blind controlled clinical trial. The experimental group received one tablet of Tenavit® daily and the placebo group received the same tablet with the organoleptic characteristics of Tenavit® for a period of 4 months. The women were assessed before the intervention and after 4 months of medication. A self-report questionnaire to assess quality of life (QSF-36) was applied and anthropometric measurements, cholesterol and fractions, triglycerides, fasting glucose, homocysteine and cysteine were evaluated. Results: The only variable that presented significant alteration in both dimensions (between and within group) was the homocysteine. It was observed statistical significant between groups in the final measure for homocysteine (control group: 11.5mmol/ L; experimental group: 9.4 mmo

DETAILED DESCRIPTION:
Subjects The study protocol and informed consent was approved by the Ethics Committee of the Hospital Santa Marcelina, Sao Paulo, Brazil (Process nº 09/08, CAAE nº 0016.0.270.000-08).Sixty women (figure 1) were postmenopausal selected from the outpatient Gynecology - Endocrine Hospital Santa Marcelina that passed by routine consultations and fulfilling the inclusion criteria were invited to the study.

Inclusion criteria were: a year of amenorrhea, FSH (follicle stimulating hormone) greater than 30mUI/ml and submit dyslipidemia, defined as LDL> 150 mg / dl15. Women with diabetes difficult to control or with recent myocardial infarction or thromboembolic diseases, severe hepatic impairment or activity were excluded. In addition, patients who had any form of cancer were excluded from the group.

Study Design The women were randomly allocated to control or experimental group (30 in each group) in a double-blind controlled clinical trial. The experimental group received one tablet of Tenavit®(pyridoxine hydrochloride 4.00mg + folic acid 0.80mg + cyanocobalamin 0.40mg) daily and the placebo group received the same tablet with the organoleptic characteristics of Tenavit® for a period of 4 months. After this period of treatment, the women were assessed.

Procedures During clinical examination, a self-report questionnaire to assess quality of life (QSF-36) that demonstrates how the individual feels regarding your activities, your health and disposition on a daily, always referring to the last month15, was applied. The Framingham Score was also applied. Framingham predictions was good in the low- to intermediate cardiovascular risk16,17.Anthropometric measurements of blood pressure, weight, height, body mass index, waist and hip were evaluated by the same medical team. Venous blood was collected on two different occasions during the study (at baseline and at end of treatment), while maintaining the 12-hour fast and the interval of 4 months between tests, both in the experimental and in the control group. Total cholesterol and fractions, triglycerides, fasting glucose, homocysteine and cysteine were performed. The dosage of plasma homocysteine and cysteine was performed by high performance liquid chromatography (HPLC).

ELIGIBILITY:
Inclusion Criteria:

* 60 women with one year of amenorrhea, FSH greater than 30, and those with dyslipidemia.

Exclusion Criteria:

* Women with difficult-to-control diabetes, recent heart attack or thromboembolic diseases, severe or active hepatic failure were excluded from this group. In addition, patients who had cancer.

Ages: 40 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-12; Primary Completion 2010-01 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
supplementation may be beneficial in postmenopausal patients, with the intention to reduce the level of homocysteine | The women were assessed before the intervention and after 4 months of medication.
  supplementation may be beneficial in postmenopausal patients, with the intention to reduce the level of homocysteine and, thus, reduce the cardiovascular risk in this age.

REFERENCES:
- [Result] Nair KG, Ashavaid TF, Nair SR, Eghlim FF. The genetic basis of hyperhomocysteinemia. Indian Heart J. 2000 Nov-Dec;52(7 Suppl):S16-17. No abstract available. PMID 11339434
- [Result] Chambers JC, McGregor A, Jean-Marie J, Obeid OA, Kooner JS. Demonstration of rapid onset vascular endothelial dysfunction after hyperhomocysteinemia: an effect reversible with vitamin C therapy. Circulation. 1999 Mar 9;99(9):1156-60. doi: 10.1161/01.cir.99.9.1156. PMID 10069782
- [Result] Nappo F, De Rosa N, Marfella R, De Lucia D, Ingrosso D, Perna AF, Farzati B, Giugliano D. Impairment of endothelial functions by acute hyperhomocysteinemia and reversal by antioxidant vitamins. JAMA. 1999 Jun 9;281(22):2113-8. doi: 10.1001/jama.281.22.2113. PMID 10367822
- [Result] Fonseca V, Guba SC, Fink LM. Hyperhomocysteinemia and the endocrine system: implications for atherosclerosis and thrombosis. Endocr Rev. 1999 Oct;20(5):738-59. doi: 10.1210/edrv.20.5.0381. No abstract available. PMID 10529901
- [Result] Lussier-Cacan S, Xhignesse M, Piolot A, Selhub J, Davignon J, Genest J Jr. Plasma total homocysteine in healthy subjects: sex-specific relation with biological traits. Am J Clin Nutr. 1996 Oct;64(4):587-93. doi: 10.1093/ajcn/64.4.587. PMID 8839504
- [Result] Selhub J, Jacques PF, Wilson PW, Rush D, Rosenberg IH. Vitamin status and intake as primary determinants of homocysteinemia in an elderly population. JAMA. 1993 Dec 8;270(22):2693-8. doi: 10.1001/jama.1993.03510220049033. PMID 8133587
- [Result] von Eckardstein A, Malinow MR, Upson B, Heinrich J, Schulte H, Schonfeld R, Kohler E, Assmann G. Effects of age, lipoproteins, and hemostatic parameters on the role of homocyst(e)inemia as a cardiovascular risk factor in men. Arterioscler Thromb. 1994 Mar;14(3):460-4. doi: 10.1161/01.atv.14.3.460. PMID 8123652
- [Result] McKinley MC. Nutritional aspects and possible pathological mechanisms of hyperhomocysteinaemia: an independent risk factor for vascular disease. Proc Nutr Soc. 2000 May;59(2):221-37. doi: 10.1017/s0029665100000252. PMID 10946791
- [Result] van Kempen BJ, Ferket BS, Kavousi M, Leening MJ, Steyerberg EW, Ikram MA, Witteman JC, Hofman A, Franco OH, Hunink MG. Performance of Framingham cardiovascular disease (CVD) predictions in the Rotterdam Study taking into account competing risks and disentangling CVD into coronary heart disease (CHD) and stroke. Int J Cardiol. 2014 Feb 15;171(3):413-8. doi: 10.1016/j.ijcard.2013.12.036. Epub 2013 Dec 27. PMID 24438922
- [Result] Gokkusu C, Ozbek Z, Tata G. Hormone replacement therapy: relation to homocysteine and prooxidant-antioxidant status in healthy postmenopausal women. Arch Gynecol Obstet. 2012 Mar;285(3):733-9. doi: 10.1007/s00404-011-2051-2. Epub 2011 Aug 30. PMID 21877144
- [Result] Reslan OM, Khalil RA. Vascular effects of estrogenic menopausal hormone therapy. Rev Recent Clin Trials. 2012 Feb;7(1):47-70. doi: 10.2174/157488712799363253. PMID 21864249
- [Result] Dodds L, Fell DB, Dooley KC, Armson BA, Allen AC, Nassar BA, Perkins S, Joseph KS. Effect of homocysteine concentration in early pregnancy on gestational hypertensive disorders and other pregnancy outcomes. Clin Chem. 2008 Feb;54(2):326-34. doi: 10.1373/clinchem.2007.097469. Epub 2007 Dec 10. PMID 18070815
- See also: Website of the Ministry of Health with mortality tables — http://tabnet.datasus.gov.br/cgi/tabcgi.exe?sim/cnv/obt10uf.def